CLINICAL TRIAL: NCT05046821
Title: Influence of NT5c1A Antibodies on Disease Progression, Clinical Phenotype and Blood and Muscle Biomarkers in Sporadic Inclusion Body Myositis - A Prospective Evaluation (INSPIRE-IBM Study)
Brief Title: Sporadic Inclusion Body Myositis Natural History Study
Acronym: INSPIRE-IBM
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Tahseen Mozaffar, Professor of Neurology, University of California, Irvine
Other Study IDs: 20216779; R01AR078340-01 (NIH)
Record Dates: First submitted 2021-09-08; First posted 2021-09-16 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Sporadic Inclusion Body Myositis; Inclusion Body Myositis
MeSH Terms: conditions — Myositis, Inclusion Body

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA and RNA will be isolated from blood and muscle samples and stored for future research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective natural history study on patients with clinically defined sIBM. Participants will be assessed every 6 months over two years (five visits total). We will include 150 participants, enrolled across 13 sites, with sporadic IBM, diagnosed according to established criteria.

DETAILED DESCRIPTION:
This is a prospective natural history study on patients with clinically defined sIBM. Participants will be assessed every 6 months over two years (five visits total). We will include 150 participants with sporadic IBM, diagnosed according to established criteria. Participants will require an routine serum sample via blood draw to evaluate for NT5c1A antibody status. This testing will be performed at Washington University School of Medicine in the Neuromuscular Laboratory. Investigators will be blinded to antibody status. A subset of participants (40) will undergo a muscle biopsy at the Baseline visit.

Aim 1. To determine for the first time whether NT5c1A antibodies mediate disease progression over a two-year interval in patients with sIBM.

We will perform a prospective, non-interventional, observational study on patients with sIBM with follow up and evaluations every 6 months over a two-year time frame. Primary analyses are: 1) the rates of disease progression and severity as measured by rates of decline in IBM Functional Rating Scale (IBMFRS) score and Timed Get Up and Go (TUG); 2) the presence or absence of serum antibodies to NT5c1A; and 3) the presence and frequency of variant T-cells in the serum and skeletal muscle.

Aim 2. To perform a detailed morphological, histochemical and immunohistochemical analysis of fresh muscle biopsy specimens obtained from a subset of patients with sIBM.

Aim 3. To characterize the distribution of "immunosenescent" lymphocytes in circulating blood from patients with sIBM.

Aim 4. To quantify the decline in the respiratory function of sIBM patients.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 40 years and older
2. Fulfills ENMC 2011 criteria of clinically definite or probable sporadic Inclusion body myositis (sIBM)
3. Disease onset is within the past 10 years of the time of Baseline visit
4. Able to participate and comply with study related procedures
5. Able to provide written consent

Exclusion Criteria:

1. Current or very recent use (within last 6 months of the Baseline visit) of immunomodulation or immunosuppression therapy.
2. Current or very recent use (within last 90 days of the Baseline visit) of an investigational medication or therapy.
3. Co-existing significant medical or surgical conditions that, in the opinion of the investigator, will influence study participation or alter natural history.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Paticipants age 40 and older with sporadic IBM, diagnosed according to established criteria.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Inclusion Body Myositis Functional Rating Scale (IBMFRS) | Change from Baseline to Month 24
  The IBMFRS is a 10 item questionnaire. Scores for each item range from 0 to 4. There is a total maximum score of 40 and minimum score of 0. The higher the score the better functional status of the person.
Timed Up and Go (TUG) | Change from Baseline to Month 24
  Stand up from a chair, walk 3 meters, sit back down in chair
Frequency of immunophenotypic abnormalities in blood and muscle | Change from Baseline to Month 24
  Laboratory assessment
Forced Vital Capacity (FVC) (sitting) | Change from Baseline to Month 24
  breathing test

SECONDARY OUTCOMES:
Manual Muscle Testing | Change from Baseline to Month 24
  muscle strength testing
Hand Held Dynamometry | Change from Baseline to Month 24
  muscle strength testing
Sydney Swallow Questionnaire | Change from Baseline to Month 24
  swallow ability questionnaire
EAT-10 Questionnaire | Change from Baseline to Month 24
  swallow ability questionnaire
NIH PROMIS questionnaires | Change from Baseline to Month 24
  quality of life questionnaires
Forced Vital Capacity (supine) | Change from Baseline to Month 24
  breathing test done while lying down
Maximum Inspiratory Pressure/Maximum Expiratory Pressure | Change from Baseline to Month 24
  breathing tests
sporadic inclusion body myositis physical functioning assessment (sIFA) | Change from Baseline to Month 24
  functional ability questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Tahseen Mozaffar, MD FAAN, FANA, Principal Investigator — University of California, Irvine
Locations (13):
- United States (13):
  - University of California, Los Angeles, Los Angeles, California
  - University of California, Irvine, Orange, California
  - University of Colorado, Aurora, Colorado
  - University of Miami, Miami, Florida
  - Kansas University Medical Center, Fairway, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Washington University in St. Louis, St Louis, Missouri
  - Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Nerve and Muscle Center of Texas, Houston, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided